CLINICAL TRIAL: NCT06800872
Title: Effect of Body Vibration Sessions on Energy Expenditure at Rest and on Cardiovascular and Musculoskeletal Parameters in Obese Boys Hospitalized for a Multidisciplinary Program of Integrated Metabolic Rehabilitation
Brief Title: Whole Body Vibration Effects on Energy Expenditure in Obese Adolescents
Acronym: VIBRAREEOB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01C413
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: Resting energy expenditure; Body vibration; Body composition; Functional tests
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): 14 boys with obesity: standard in-hospital protocol of multidisciplinary metabolic rehabilitation
  Interventions: Other: Multidisciplinary metabolic rehabilitation
- Experimental group (Experimental): 14 boys with obesity: standard in-hospital protocol of multidisciplinary metabolic rehabilitation + 24 sessions (2 sessions per day) of 30 minutes each of training on a vibration platform.
  Interventions: Other: Multidisciplinary metabolic rehabilitation + training with WBVE

INTERVENTIONS:
Other: Multidisciplinary metabolic rehabilitation — Standard in-hospital protocol of multidisciplinary metabolic rehabilitation
  Arms: Control group
Other: Multidisciplinary metabolic rehabilitation + training with WBVE — Standard in-hospital protocol of multidisciplinary metabolic rehabilitation + 24 sessions (2 sessions per day) of 30 minutes each of training on a vibration platform (WBVE)
  Arms: Experimental group

SUMMARY:
The main aim of the present study is to evaluate in a group of adolescents with obesity, hospitalized for a period of integrated metabolic rehabilitation (calorie restriction, aerobic physical activity, psychological counseling, nutritional re-education) lasting 3 weeks, the effects produced from a period of training with vibration stimulation on vibration platforms (Whole Body Vibration Exercise [WBVE]) on the resting energy expenditure (REE), assessed through indirect calorimetry. The results will be compared with those obtained in a control group, subjected to integrated metabolic rehabilitation alone.

Secondary aims of the study are to evaluate the effects of training with WBVE also on cardiovascular and musculoskeletal parameters, evaluated through specific functional tests, comparing them with those obtained in the control group.

DETAILED DESCRIPTION:
The main aim of the present study is to evaluate in a group of adolescents with obesity, hospitalized for a period of integrated metabolic rehabilitation (calorie restriction, aerobic physical activity, psychological counseling, nutritional re-education) lasting 3 weeks, the effects produced from a period of training with vibration stimulation on vibration platforms (Whole Body Vibration Exercise [WBVE]) on the resting energy expenditure (REE), assessed through indirect calorimetry. The results will be compared with those obtained in a control group, subjected to integrated metabolic rehabilitation alone.

Secondary aims of the study are to evaluate the effects of training with WBVE also on cardiovascular and musculoskeletal parameters, evaluated through specific functional tests, comparing them with those obtained in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age range 13-18 years
* Obesity (Body Mass Index Standard Deviation Score > 2)
* Hospitalization for a multidisciplinary program of integrated metabolic rehabilitation at the Division of Auxology, S. Giuseppe Hospital, Istituto Auxologico Italiano, IRCCS, Piancavallo, Italy

Exclusion Criteria:

* Presence of cardiovascular, psychiatric, and musculoskeletal pathologies
* Absence of signed written consent

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Resting energy expenditure | At baseline and after 3 weeks
  Resting energy expenditure assessed through indirect calorimetry.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy